CLINICAL TRIAL: NCT00949416
Title: Risk Factors of Incidence of Type 2 Diabetes and Cardiovascular Diseases
Brief Title: Risk Factors of Incidence of Type 2 Diabetes and Cardiovascular Diseases---Shanghai Baoshan Study
Acronym: SBSS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Ruijin Hospital, Shanghai Jiaotong University School of Medicine
Other Study IDs: CCEMD007
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes; Cardiovascular Disease
Keywords: genetic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective: Recruit 3 cohorts with 1000-1200 subjects each: people with normal glucose metabolism, impaired glucose regulation (IGR), and with Type 2 diabetes. To study the risk factors in development of type 2 diabetes.

DETAILED DESCRIPTION:
Methods:

We aim to perform a two-step blood glucose survey in 2008-2009 in a population selected from a single urban community of Shanghai. The Institutional Review Board of the Rui-Jin Hospital approved the study protocol. Informed consent will be obtained from each participant.

1. In the first step, we first invited all registered permanent residents aged 40 or above by local poster advertisement and by mail to participate in a screening examination, during which we collected information on lifestyle, medical history and the use of medications using a questionnaire, and performed anthropometrical measurements and fasting glucose measurement. The first step of diabetes screening finished in June, 2008.
2. In the second step, after exclusion of subjects with self-reported diabetes, we classified the screened subjects into 3 groups according to their fasting plasma glucose concentration of 7.0 mmol/L or above, 5.0 to 6.9 mmol/L or below 5.0 mmol/L. We selected randomly a sample from these 3 subgroups for further investigation including a 75-g oral glucose tolerance test (OGTT) and blood and urine sampling and other vascular functional measurements. Our selection was based on a ratio of 1:1.2:1.44, because of the concern that by knowing the results of fasting plasma glucose test, subjects with lower glucose levels might have a lower participation rate than those with higher glucose concentrations. Nevertheless, this ratio was arbitrarily chosen. Finally, 1000 Type 2 diabetic patients, 1200 subjects with IGR and 1440 subjects with normal glucose metabolism were selected as target population of this study by random sampling for further blood and urine sampling.
3. Biomarkers and genetic risk factors will be evaluated in the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* aged above 40 years

Exclusion Criteria:

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 Type 2 diabetic patients, 1200 subjects with IGR and 1440 subjects with normal glucose metabolism (aged above 40 years old, both men and women)were selected as target population of this study by random sampling.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD, PHD, Study Chair — Shanghai Clinical Centre for Endocrinology and Metabolism